CLINICAL TRIAL: NCT06507709
Title: Radiographic Changes in the Maxillary Sinus Following Closed Sinus Augmentation With Calcium Phosphosilicate
Brief Title: Closed Sinus Augmentation With a Calcium Phosphosilicate Putty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00000739
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant; Maxillary Sinus Floor Augmentation
Keywords: Cone beam computed tomography; Calcium Phosphosilicate putty

STUDY DESIGN:
Intervention Model Description: Case series single group with no control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed sinus augmentation with Calcium Phosphosilicate Putty (Experimental): Use of CBCT immediately post-operatively after placement of Calcium Phosphosilicate Putty used as standard of care for closed sinus augmentation and at 6 months after surgery.
  Interventions: Procedure: Low volume CBCT

INTERVENTIONS:
Procedure: Low volume CBCT — 3-D imaging used during dental practice
  Other Names: Cone Beam Computed Tomography

SUMMARY:
The goal of this clinical study is to learn if cone beam computed tomography (CBCT) or 3-dimensional x-ray can help to let the investigator know if dental implant placement can be done after performing closed sinus surgery.

The study will look at the structure of your gum where the implant will be placed after performing the surgery using 3-D x-ray and compare that to how the structure of your gum looks 6 months later.

The 3-D imaging will happen after standard of care surgery to prepare your gum for an implant and then 6 months later to verify that the site is ready for the implant.

DETAILED DESCRIPTION:
While you are taking part in this study, participants will be asked to attend approximately two visits with the researchers or study staff. For research purposes, one visit is the surgical appointment and a postoperative visit at six months, these will likely be scheduled at standard of care visits.

If the participant elects a dental implant for tooth replacement, your sinus grafting will be performed, and the dental implant will be placed on the same appointment.

Study Procedures - as a participant in this research, you will undergo the following procedures:

1. Immediately upon completion of your sinus grafting and dental implant placement a three-dimensional x-ray will be taken in the Graduate Periodontics clinic.
2. At six months following your dental implant placement an additional three-dimensional x-ray will be taken in the Graduate Periodontics clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant to understand and the willingness to sign a written informed consent document.
2. English speaking.
3. Individuals who are normal healthy or have a diabetes diagnosis with a current HbA1c (glycated glucose)< 7.0.
4. Partially edentulous patients (18-85 years of age) requiring maxillary sinus augmentation for dental implant placement
5. At minimum 5mm of native bone below the maxillary sinus inferior border

Exclusion Criteria:

1. Maxillary sinus disease
2. Diabetes diagnosis with a current HbA1c > 7.1 or greater due to diabetes effect on bone metabolism
3. Pregnant or attempting to become pregnant
4. Having a disease that affects bone metabolism
5. Use of medications known to affect bone metabolism
6. Tobacco, cannabis or vaping use
7. Alcoholism or other recreational drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Bone Volume change | Baseline to 6 months
  Bone volume changes will be reported as a percentage, with mean, median, and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Powell, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be thoroughly de-identified and will not be traceable to a specific study participant. Data will be shared through publication in a peer review journal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available in a journal at study end at the time of publication.